CLINICAL TRIAL: NCT04066023
Title: Randomized, Double-Blind, Multi-Center, Parallel-Group Comparison of the Efficacy and Safety of the C213 (Zolmitriptan Microneedle System) to Placebo for the Acute Treatment of Cluster Headaches
Brief Title: Double-Blind Comparison of the Efficacy and Safety of C213 to Placebo for the Acute Treatment of Cluster Headaches
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-2019-001
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Cluster Headache
Keywords: Episodic cluster headache; Chronic cluster headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Intervention Model Description: Qualified subjects are assigned to received a single administration of one of three blinded treatment assignments (one of two dose levels or placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, care providers, investigator, and outcomes assessors are blinded to randomized treatment assignment. Study drugs are blinded and identical in appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- C213 1.9 mg (Experimental): C213, 1.9 mg administered as one 1.9 mg patch and one placebo patch
  Interventions: Drug: C213 Microneedle System
- C213 3.8mg (Experimental): C213 3.8 mg administered as two 1.9 mg patches
  Interventions: Drug: C213 Microneedle System
- Placebo (Placebo Comparator): Placebo microneedle system administered as two placebo patches
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C213 Microneedle System — The C213 System is a proprietary disposable patch and a reusable applicator. The zolmitriptan-coated titanium microneedle array (3 cm^2 array) is attached to a 5 cm^2 adhesive patch.
  Other Names: Zolmitriptan Microneedle System
  Arms: C213 1.9 mg; C213 3.8mg
Drug: Placebo — The C213 System is a proprietary disposable patch and a reusable applicator. The placebo patch is a single use, 3 cm^2 Placebo (intracutaneous microneedle) system that contains no active ingredients.
  Other Names: ZP Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled study. Subjects who meet the entry criteria will be randomized o receive one of three blinded treatments [C213 1.9 mg patch and placebo patch; C213 3.8 mg (1.9 mg x 2 patches), two placebo patches] on Day 1 and will have up to 48 weeks to confirm and treat a cluster headache. Subjects will self-administer the patches and respond to questions in the electronic diary (eDiary) until 1-hour post treatment administration.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study. Approximately 120 subjects who meet the entry criteria will be randomized 1:1:1 to receive one of three blinded treatments [C213 1.9 mg patch and placebo patch; C213 3.8 mg (1.9 mg x 2 patches), two placebo patches].

Qualified subjects will randomize to the double-blind treatment period at Day 1 and will have up to 48 weeks to confirm and treat a cluster headache. Using the eDiary to confirm they are experiencing a cluster headache, subjects will self-administer the patches and continue to respond to questions in the eDiary until 1-hour post treatment administration.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. Women or men 18 to 65 years of age
3. Greater than 1-year history of episodic or chronic cluster headache with onset prior to 50 years of age. Diagnosis must comply with ICHD-3 (International Headache Society (IHS) diagnostic criteria). Diagnostic criteria must include a history of at least 5 attacks not attributed to any other disorder that include all of the following criteria:

   1. Severe or very severe unilateral orbital, supraorbital and/or temporal pain lasting 45-180 minutes (average, when untreated)
   2. Either or both of the following:

      1. At least one of the following symptoms or signs, ipsilateral to the pain:

         1. Conjunctival injection and/or lacrimation
         2. Nasal congestion and/or rhinorrhea
         3. Eyelid edema
         4. Forehead and facial sweating
         5. Miosis and or/ptosis
      2. A sense of restlessness or agitation
   3. Attacks have a frequency between one every other day and eight per day for more than half of the time when the disorder is active.
   4. Not better accounted for by another International Classification of Headache Disorders (ICHD) diagnosis
4. Cluster history during the 12-month period prior to the screening visit must include:

   1. At least 1 cluster period
   2. Averaging 2-6 headaches per day
   3. Lasting at least 7 days
5. Subject can distinguish cluster headaches from other headaches (i.e., migraine and tension-type headaches)
6. Women of child-bearing potential must not be pregnant, must agree to avoid pregnancy during the trial, and must use one of the following or be surgically sterilized: intrauterine device, or a hormonal contraceptive
7. Able to understand the operation of the electronic diary and able to apply the demo study drug patch correctly.

Exclusion Criteria:

1. Contraindications to triptans
2. Use of any prohibited concomitant medications within 30 days of screening
3. History of hemiplegic migraine or migraine with brainstem aura
4. Participation in another investigational trial within 30 days or 5 half-lives of investigational product (whichever is longer).
5. Previous M207/C213 exposure in a clinical trial
6. Subject has other significant pain problems that might confound the study assessments in the opinion of the investigator
7. Diagnosis of any malignant disease (other than adequately treated or excised non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin) within the 5 years prior to screening
8. History of unstable psychiatric illness requiring medication or hospitalization in the 12 months prior to study initiation
9. Subjects who have a known allergy or sensitivity to zolmitriptan or its derivatives or formulations
10. Subjects who have a known allergy or sensitivity to adhesions
11. Subjects who have skin lesions or tattoos covering the entire potential area(s) of C213 application
12. Woman who are pregnant, breast-feeding or plan a pregnancy during this study
13. Clinically significant liver disease [Alanine Aminotransferase (ALT) > 150 U/L; Aspartate Aminotransferase (AST) > 130 U/L or bilirubin > 2x ULN]
14. Clinically significant kidney disease (eGFR < 60 ml/min / 1.73 m² or to creatinine > 1.5 x ULN)
15. Subject has clinically significant ECG findings, defined by:

    1. ischemic changes (defined as > 1mm of down-sloping ST segment depression in at least two contiguous leads)
    2. Q-waves in at least two contiguous leads
    3. clinically significant intra-ventricular conduction abnormalities (left bundle branch block or Wolf-Parkinson-White syndrome)
    4. clinically significant arrhythmias (e.g., current atrial fibrillation)
16. History of coronary artery disease (CAD), coronary vasospasm (including Prinzmetal's angina), aortic aneurysm, peripheral vascular disease or other ischemic diseases (e.g., ischemic bowel syndrome or Raynaud's syndrome)
17. Three or more of the following CAD risk factors:

    1. Current tobacco use
    2. Hypertension (systolic BP > 140 or diastolic BP > 90) or receiving anti-hypertensive medication for treatment of hypertension
    3. Hyperlipidemia - LDL > 159 mg/dL and/or HDL < 40 mg/dL (or on prescribed anti-cholesterol treatment)
    4. Family history of premature coronary artery disease (CAD) (< 55 years of age in male first-degree relatives or < 65 years of age in female first degree relatives)
    5. Diabetes mellitus
18. History of cerebral vascular accident (CVA), transient ischemic attacks (TIA), or seizures
19. History of concurrent illness that requires hospitalization within 30 days prior to study initiation
20. Any other household member currently participating in a C213 study or relative of site staff member
21. Any reason to believe that compliance with the study requirements and completion of evaluations required for this study will not be possible
22. Any language barrier that, in the opinion of the Investigator, would preclude communication and compliance with the study requirements
23. History or current abuse of or dependence on alcohol or drugs that would interfere with the results or adherence to study requirements
24. Any positive drug screens for phencyclidine (PCP), 3,4-methylenedioxy-methamphetamine (MDMA) (ecstasy), cocaine, and/or meth/amphetamine(s)
25. Current or planned use of hallucinogens (e.g. psilocybin) during the trial
26. Any clinically relevant abnormal findings in the physical exam, vital signs or laboratory tests that, in the opinion of the Investigator, may put the subject at risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Kellerman, PharmD, Study Director — Zosano Pharma Corporation
Locations (12):
- United States (12):
  - Keck Medicine of USC, Los Angeles, California
  - Stanford University, Palo Alto, California
  - California Medical Clinic for Headache, Santa Monica, California
  - KI Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - Atlanta Headache Specialists, Atlanta, Georgia
  - New England Regional Headache Center, Inc., Worcester, Massachusetts
  - Nevada Headache Institute, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dent Neuro Institute, Buffalo, Amherst, New York
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center- Neurology Clinic, Dallas, Texas
  - Medstar Georgetown University Hospital at McLean, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 subjects were screened at 12 investigative sites. Of the 51 screened subjects, 42 were randomized to receive either C213 1.9 mg (17 subjects), C213 3.8 mg (13), or placebo (12) and had up to 48 weeks from randomization to treat a qualifying headache. 23 subjects applied the study patch and entered the Treatment Period.
Period: Overall Study
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Started | 12 | 17 | 13
Completed | 9 | 9 | 7
Not Completed | 3 | 8 | 6
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Sponsor decision | 3 | 6 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Noncompliance | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg | Total
Number analyzed (Participants) | 9 | 9 | 5 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (11.82) | 50.3 (12.75) | 45.4 (12.76) | 50.1 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 8 | 6 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 8 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 9 | 8 | 3 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 5 | 23
Weight [Mean (Standard Deviation); unit: kilograms] | 94.9 (9.76) | 85.3 (13.36) | 82.6 (14.88) | 88.4 (12.98)
Height [Mean (Standard Deviation); unit: centimeters] | 180.0 (8.92) | 174.3 (9.14) | 173.7 (7.53) | 176.5 (8.82)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (3.51) | 28.4 (4.54) | 27.2 (3.27) | 28.6 (3.79)
Nicotine User [Count of Participants; unit: Participants]
  Never | 3 | 4 | 2 | 9
  Past | 2 | 3 | 2 | 7
  Current | 4 | 2 | 1 | 7
Current Alcohol User [Count of Participants; unit: Participants] | 5 | 3 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieve Pain Relief
Description: Pain relief is defined by a decrease in pain from severe to mild or none without the use of acute rescue medication.
Time Frame: 15 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 3 | 5 | 5

2. Primary Outcome: Percentage of Subjects Who Achieve Sustained Pain Relief
Description: Sustained pain relief requires a pain rating of mild or none at each timepoint from 15 minutes to 60 minutes without the use of acute rescue medication.
Time Frame: 15 minutes to 60 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 3 | 4 | 5

3. Secondary Outcome: Percentage of Subjects That Achieve Pain Relief
Description: Pain relief is defined by a decrease in pain from severe to mild or none without the use of acute rescue medication.
Time Frame: 5 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 0 | 2 | 1

4. Secondary Outcome: Percentage of Subjects That Achieve Sustained Pain Relief
Description: Sustained pain relief requires a pain rating of mild or none at each timepoint within the time frame without the use of acute rescue medication.
Time Frame: 5 minutes to 60 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 0 | 2 | 1

5. Secondary Outcome: Percentage of Subjects That Achieve Pain Freedom
Description: Pain freedom is defined by a decrease in pain from severe to none without the use of acute rescue medication.
Time Frame: 10 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 0 | 1 | 1

6. Secondary Outcome: Percentage of Subjects That Achieve Sustained Pain Freedom
Description: Sustained pain freedom requires a pain rating of none at each timepoint within the time frame without the use of acute rescue medication.
Time Frame: 15 to 60 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 1 | 2 | 2

7. Secondary Outcome: Percentage of Subjects Able to Perform Their Usual Daily Activities as Assessed by the Subject
Description: Whether or not subjects were able to perform their usual daily activities was assessed by subject responses (Yes or No) in the electronic diary (eDiary) to the question, "Do you feel able to perform your usual daily activities?" If a subject responded "Yes" but had used a rescue medication, the subject was considered as not being able to perform the usual daily activities.
Time Frame: within 20 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 2 | 5 | 4

8. Secondary Outcome: Percentage of Subjects That Achieve Pain Relief
Description: Pain relief is defined by a decrease in pain from severe to mild or none without the use of acute rescue medication
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 2 | 3 | 3

9. Secondary Outcome: Percentage of Subjects That Achieve Pain Relief
Description: Pain relief is defined by a decrease in pain from severe to mild or none without the use of acute rescue medication.
Time Frame: 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 4 | 5 | 4

10. Secondary Outcome: Percentage of Subjects That Achieve Sustained Pain Relief
Description: as for outcome 4
Time Frame: 10 minutes to 60 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 2 | 3 | 3

11. Secondary Outcome: Percentage of Subjects That Achieve Pain Freedom
Description: Pain freedom is defined by a decrease in pain from severe to none without the use of acute rescue medication.
Time Frame: 20 minutes
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
Number analyzed (Participants) | 8 | 9 | 5
Participants | 2 | 3 | 3

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were collected for 8 days (+3 days) from patch application through the End of Study or Early Discontinuation visit, up to 48 weeks
Arm/Group | Placebo | C213 1.9 mg | C213 3.8mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 1/9 | 4/9 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | C213 1.9 mg (N=9) | C213 3.8mg (N=7)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Mild skin erythema from sunburn on right and left upper arms
Application site erythema (General disorders) | 1 (1) | 2 (2) | 0 (0) — Application site--mild erythema on right upper arm
Application site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) — Application site--mild skin edema right upper arm
Application site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) — Left arm application site bruising
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Coronavirus subject tested positive and was asymptomatic
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Tonsillitis
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — First degree atrioventricular block

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic had significant impact: Enrollment was hampered; therefore, Zosano ended the trial with 42 subjects randomized and 23 subjects who treated a Cluster attack. The study was thus underpowered to detect a difference between C213 doses and placebo. The protocol was amended to allow for feasible assessments to be done virtually and permit in home monthly pregnancy testing. The monitoring plan and Zosano Pharma vendor management plan were updated to allow for remote monitoring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04066023/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT04066023/SAP_001.pdf